CLINICAL TRIAL: NCT07012512
Title: Adjusted Study Protocol: Within-Subject Paired-Eye Design Comparing Pilocarpine 0.1%, Phentolamine 0.75%, and Combination Therapy for Cyclopentolate Reversal in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Mansoura university Ophthalmic
Record Dates: First submitted 2025-05-30; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Pupillary Constriction; Accomodation
MeSH Terms: conditions — Miosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilocarpine group (Experimental): Children will receive pilocarpine drops in one eye and placebo in the other
  Interventions: Drug: Pilocarpine 0.1%
- Phentolamine group (Active Comparator): Children will receive phentolamine eye drop in one eye and placebo in the other
  Interventions: Drug: Use of phentolamine eye drops to reverse cycloplegia
- Combined (Experimental): Children will receive a combination of pilocarpine and placebo in one eye and placebo in the other
  Interventions: Drug: Combination of pilocarpine 0.1% and phentolamine 0.75%

INTERVENTIONS:
Drug: Use of phentolamine eye drops to reverse cycloplegia — Use of phentolamine 0.75% eye drops to reverse cycloplegia
  Arms: Phentolamine group
Drug: Pilocarpine 0.1% — Use of pilocarpine 0.1% to reverse cycloplegia
  Arms: Pilocarpine group
Drug: Combination of pilocarpine 0.1% and phentolamine 0.75% — Combination of pilocarpine 0.1% and phentolamine 0.75%
  Arms: Combined

SUMMARY:
The study aims at reversing pupillary dilatation. and cycloplegia in children undergoing cycloplegic refraction for eyeglasses prescription and ocular examination. This will be achieved using pilocarpine , phentolamine or a combination. This may help decrease the glare and improve near vision early to decrease unwanted effects of cycloplegic drops.

DETAILED DESCRIPTION:
To compare the efficacy of pilocarpine 0.1%, phentolamine 0.75%, and combined therapy in reversing cyclopentolate-induced cycloplegia/mydriasis in pediatric patients using a within-subject paired-eye design (treated vs. untreated eye).

Interventions

Cycloplegia Induction:

Both eyes receive cyclopentolate 1% (2 drops, 5 minutes apart). Then cycloplegic effect confirmed at 30 minutes (accommodation ≤2 D, pupil ≥6 mm).

Reversal Agents (administered at 30 minutes post-cyclopentolate):

Pilocarpine group: Pilocarpine 0.1% (1 drop) in the study eye; placebo in the control eye.

Phentolamine group: Phentolamine 0.75% (1 drop) in the study eye; placebo in the control eye.

Combination: Pilocarpine 0.1% + phentolamine 0.75% (1 drop each) in the study eye; placebo in the control eye.

ELIGIBILITY:
Inclusion Criteria:

* Children between 5 and 12 years undergoing cycloplegia

Exclusion Criteria:

* Patient refusal

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Reversal of pupillary dilatation | Hourly for four hours after administration of the drug

SECONDARY OUTCOMES:
Recovery of accommodation after instillation of the drop | Hourly for four hours after administration of the drug

IPD SHARING:
Plan to Share IPD: No